CLINICAL TRIAL: NCT03183570
Title: Detection of Integrin avb6 in Idiopathic Pulmonary Fibrosis, Primary Sclerosing Cholangitis, and Coronavirus Disease 2019 With [18F]FP-R01-MG-F2 With PET/CT
Brief Title: Detection of Integrin avb6 in IPF, PSC, and COVID19 Using PET/CT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Haiwei Henry Guo, Clinical Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB Protocol: 40450
Record Dates: First submitted 2017-05-08; First posted 2017-06-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Primary Sclerosing Cholangitis; Covid19 Pneumonia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- [18F]FP-R01-MG-F2 PET/CT in IPF Patients, Recovered COVID19 Patients, and Healthy Volunteers (Experimental): Arm1: 7mCi (range 6-9 mCi) [18F]FP-R01-MG-F2 will be administered to the study participant. A 60-minute dynamic PET/CT scan to the center of the lungs in the FOV is followed by two vertex-to-thigh PET/CT scans.
  NOTE: If the patient cannot tolerate lying down for an extended period of time at the time of imaging, the patient may be switched to scanning protocol Option B, which does not include an initial 60-minute dynamic PET/CT scan.
  IPF Patients will have a repeat [18F]FP-R01-MG-F2 PET/CT scan performed within 3-8 weeks post initial scan (within 12-24 months post initial scan for previously scanned IPF patients if they are willing to be re-consented).
  Interventions: Drug: [18F]FP-R01-MG-F2
- [18F]FP-R01-MG-F2 PET/CT in PSC Patients (Experimental): Arm 2: 7mCi (range 6-9 mCi) [18F]FP-R01-MG-F2 will be administered to the study participant. A 60-minute dynamic PET/CT scan to the center of the liver in the FOV is followed by two vertex-to-thigh PET/CT scans.
  Patients will have the option for a repeat [18F]FP-R01-MG-F2 PET/CT scan performed within 3-8 weeks post initial scan.
  Interventions: Drug: [18F]FP-R01-MG-F2
- [18F]FP-R01-MG-F2 PET/CT in actively infected COVID19 Patients (Experimental): Arm 3: 7mCi (range 6-9 mCi) [18F]FP-R01-MG-F2 will be administered to the study participant. One vertex-to-thigh PET/CT scans to the center of the lung in the FOV will follow approximately 60 min post-injection.
  Interventions: Drug: [18F]FP-R01-MG-F2

INTERVENTIONS:
Drug: [18F]FP-R01-MG-F2 — 7mCi (range 6-9mCi) [18F]FP-R01-MG-F2 will be administered

SUMMARY:
Detection of Integrin avb6 in Idiopathic Pulmonary Fibrosis, Primary Sclerosing Cholangitis, and Coronavirus Disease 2019 with [18F]FP-R01-MG-F2 with PET/CT

DETAILED DESCRIPTION:
Stanford University has developed a new PET tracer, [18F]FP-R01-MG-F2, that selectively binds to integrin avb6, a cell surface receptor that is overexpressed in idiopathic pulmonary fibrosis (IPF). Increased avb6 receptors on IPF lung tissue has been well documented, while its expression remains relatively non-existent in the healthy adult lung.

The PET tracer's application will be expanded in primary sclerosing cholangitis (PSC) and COVID-19 pneumonia. The integrin avb6 is also up-regulated in the biliary epithelial cells, which drive the progression of biliary tree strictures and liver fibrosis through activation of TGF-b, as shown in IPF. Similarly, COVID-19 pneumonia is caused by the SARS-CoV-2 and leads to acute lung injury and integrin avb6 up-regulation.

The selected PET tracer [18F]FP-R01-MG-F2 has shown promise in identifying integrin avb6 in both preclinical and clinical studies at Stanford University. The investigators have demonstrated low [18F]FP-R01-MG-F2 radiopharmaceutical uptake in the heart and lung region of healthy volunteers, which was an expected biodistribution (the normal tissue uptake of the radiopharmaceutical within the body) based on immunohistochemical staining of healthy lung tissue, which demonstrated the presence of minimal avb6 receptors in healthy lung tissue.

OBJECTIVE:

1. Exploring the use of the investigational radiopharmaceutical [18]FFP-R01-MG-F2 as a biomarker for avb6 integrin in fibrotic lung tissue.
2. Exploring the use of the investigational radiopharmaceutical [18]FFP-R01-MG-F2 to access inflammation and fibrosis in the bile duct and liver.
3. Exploring the use of the investigational radiopharmaceutical [18]FFP-R01-MG-F2 to assess lung injury in COVID-19 pneumonia.

The performance of [18F]FP-R01-MG-F2 PET/CT will be assessed in a cohort of up to 13-15 IPF patients, 5 PSC patients, 5 COVID19 pneumonia patients, and 5 age-matched healthy controls. Feasibility will be measured by drawing regions of interest (ROI) around the lung/ liver of participants with IPF, COVID19, or PSC, respectively, and the lungs of healthy adult volunteers and comparing the calculated standardized uptake value maximum(s) (SUV max).

The tracer's biodistribution, safety, and tolerability will also be studied.

Recruitment of IPF subjects and healthy volunteers has been completed, although recruitment for other aspects of this clinical trial is ongoing.

ELIGIBILITY:
1.0 Eligibility Criteria for IPF Patients

1.1 Inclusion Criteria

The following inclusion criteria will be monitored:

* Patient is >/= 18 years old
* Patient is capable of making an informed decision regarding his/her treatment
* Patient diagnosed with IPF by a pulmonologist according to ATS guidelines
* Patient has high-resolution CT with definite Usual Interstitial Pneumonia (UIP) pattern
* Patient has PFT's within the last 12 months with:

  * FVC<85% predicted
  * DLCO<65% predicted
* FEV1/FCV ratio >70%
* Patient is able to comply with study procedures

  * Scanning Option A OR
  * Scanning Option B

1.2 Exclusion Criteria

The following exclusion criteria will be monitored:

* Patient with a serious uncontrolled concurrent medical illness that would limit compliance with study requirements
* Patient has a history of any clinically significant lung disease other than IPF as determined by a pulmonologist
* Patient has had a lung infection of any kind in the last 3 months
* Patient is pregnant or lactating

2.0 Eligibility Criteria for PSC Patients

2.1 Inclusion Criteria

The following inclusion criteria will be monitored:

* Patient is >/= 18 years old
* Patient is capable of making an informed decision regarding his/her treatment
* Patient diagnosed with large duct PSC, based on an abnormal cholangiography as assessed by magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography (ERCP), and/or percutaneous transhepatic cholangiopancreatography (PTC) in the context of cholestatic liver chemistry
* Patient is able to comply with study procedures

  * Scanning Option C

2.2 Exclusion Criteria

The following exclusion criteria will be monitored:

* Patient with a serious uncontrolled concurrent medical illness that would limit compliance with study requirements
* Patient has other causes of liver disease, including secondary sclerosing cholangitis or viral, metabolic, or alcoholic liver disease, as assessed clinically
* Patient has a history of ascending cholangitis within 60 days of screening, as assessed clinically
* Patient has history, current clinical or radiological suspicion, or diagnosis of cholangiocarcinoma, other hepatobiliary malignancy, colorectal cancer, or other abdominal malignancy at any time
* Presence of a percutaneous drain or bile duct stent
* Patient is pregnant or lactating

3.0 Eligibility Criteria for Healthy Controls

3.1 Inclusion Criteria

The following inclusion criteria will be monitored:

* Person is >/= 45 years old
* Person is capable of making an informed decision regarding his/her treatment
* Person is able to comply with study procedures

  * Scanning Option A OR
  * Scanning Option B

3.2 Exclusion Criteria

The following exclusion criteria will be monitored:

* Person with a serious uncontrolled concurrent medical illness that would limit compliance with study requirements
* Person has a history of any clinically significant lung disease other than IPF as determined by a pulmonologist
* Person had lung infection of any kind in the last 3 months
* Person is pregnant or lactating

4.0 Eligibility Criteria for COVID-19 patients

4.1 Inclusion Criteria

The following inclusion criteria will be monitored:

* Patient is >/= 18 years old
* Patient is capable of making an informed decision regarding his/her treatment
* Patient with a history of SARS-CoV-2 (active or recovered) infection, based on positive RT-PCR testing
* Recovered COVID-19 patient must show evidence of being non-infectious (per Stanford guideline):

  * Symptomatic, non-immunocompromised outpatients are considered COVID neg after 10 days or 3 days after symptoms resolve, whichever is longer.
  * Severely symptomatic or is immunocompromised outpatients are considered non-infectious after 20 days.
  * or RT-PCR negative x2, spaced >24 hrs apart
* Patient shows or has shown evidence of pulmonary opacities as visualized on chest radiograph or CT
* Patient is able to comply with study procedures and infection control instructions

  * Recovered COVID 19 patients: Scanning Option A OR
  * Recovered COVID-19 patients: Scanning Option B
  * COVID-19 patients with active infection or no evidence of non-active infection: Scanning Option D

4.2 Exclusion Criteria

The following exclusion criteria will be monitored:

* Person with serious uncontrolled concurrent medical illness, such as severe hypoxia, that would limit compliance with study and infection control requirements
* Person with pre-existing fibrosing lung disease (such as but not limited to IPF, NSIP, HP, and sarcoidosis prior to COVID-19 infection).
* Person is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
SUV max comparison : IPF versus Healthy Lung, PSC versus Healthy Liver, COVID19 versus Healthy Lung | an estimated average of 2 hours
  The SUVmax in a lung or liver with known IPF, COVID19 pneumonia, or PSC respectively will be compared to the SUVmax in a known healthy lung/liver. It is expected that the SUV max, which is a measurement of the maximum value of radiopharmaceutical uptake within the region of interest (ROI) in IPF, COVID19 pneumonia, and PSC will be higher than the SUV max in the healthy lung/liver.

SECONDARY OUTCOMES:
Time Activity Measurements | an estimated average of 1 hours
  Blood samples for blood time-activity measurements taken at 1, 3, 5, 10, 30, and 60 minutes after tracer injection for tracer kinetic analysis. Tracer kinetic analysis shows radiopharmaceutical distribution from the blood to the tissues over time.
Incidence of Study Completion (Safety and Tolerability) | an estimated average of 2 hours
  Vital signs and laboratory data collected before IV injection of [18F]FP-R01-MG-F2 and after completion of the scan will allow the investigators to evaluate the safety and tolerability of the radiopharmaceutical. This will be measured as the number of patients who successfully completed the study.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Guo, MD, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kimura RH, Wang L, Shen B, Huo L, Tummers W, Filipp FV, Guo HH, Haywood T, Abou-Elkacem L, Baratto L, Habte F, Devulapally R, Witney TH, Cheng Y, Tikole S, Chakraborti S, Nix J, Bonagura CA, Hatami N, Mooney JJ, Desai T, Turner S, Gaster RS, Otte A, Visser BC, Poultsides GA, Norton J, Park W, Stolowitz M, Lau K, Yang E, Natarajan A, Ilovich O, Srinivas S, Srinivasan A, Paulmurugan R, Willmann J, Chin FT, Cheng Z, Iagaru A, Li F, Gambhir SS. Evaluation of integrin alphavbeta6 cystine knot PET tracers to detect cancer and idiopathic pulmonary fibrosis. Nat Commun. 2019 Oct 14;10(1):4673. doi: 10.1038/s41467-019-11863-w. PMID 31611594
- See also: Related Info — https://doi.org/10.1038/s41467-019-11863-w